CLINICAL TRIAL: NCT03972007
Title: Effect of Light-emitting Diode (LED) Photobiomodulation Therapy on Muscular Fatigue in University Handball Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, Director, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Photobiomodulation on Strength
Record Dates: First submitted 2019-05-27; First posted 2019-06-03 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Muscular Injury
Keywords: Physiotherapy; Muscle resistance; LED; Athletic performance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Immediate LEDT Group (Experimental): The 940nm LED blanket will be positioned across the full length of the biceps brachii muscle in the dominant limb immediately before the muscle fatigue protocol.
  Interventions: Device: Fotobiomodulation
- LEDT Group 15Min (Experimental): The 940nm LED blanket will be positioned across the length of the biceps brachii muscle in the dominant limb 15 minutes before the muscle fatigue protocol.
  Interventions: Device: Fotobiomodulation
- Immediate Sham Group (Sham Comparator): The 940nm LED blanket will be positioned throughout the biceps brachii muscle in the dominant limb, however, it will not be ligated, with no light emission, immediately prior to the muscle fatigue protocol.
  Interventions: Device: Fotobiomodulation
- Sham Group 15Min (Sham Comparator): The 940nm LED blanket will be positioned throughout the biceps brachii muscle in the dominant limb, however, it will not be ligated, with no light emission, 15 minutes before the protocol of muscle fatigue.
  Interventions: Device: Fotobiomodulation

INTERVENTIONS:
Device: Fotobiomodulation — A 16x28 cm LED blanket containing 160 LEDs will be used and will use a total energy per area of 60J, with a wavelength of 940nm, just before the muscle fatigue protocol and will be applied throughout the Biceps extension.

SUMMARY:
Introduction: Low-intensity laser therapy (LBI) is a therapeutic modality with a large number of clinical studies in recent years, taking into account its effectiveness in tissue repair, pain control and, more recently, to increase performance. It is known that LED therapy has immediate effects. Therefore, analyzing the TLED in the infrared spectrum for acute responses at different times along with fatigue resistance capabilities, heart rate variability and biochemical response to fatigue in handball athletes becomes necessary. Objective: To analyze the acute effects of LED phototherapy (940nm) on fatigue resistance and recovery after strenuous exercises of university athletes. Method: The study sample will consist of 32 and 36 male athletes, for biceps brachii and quadriceps femoris, respectively. The athletes will be randomly assigned into four groups: Immediate TLED (TLED-I), TLED 15Min (TLED-15), Immediate Sham (Sham-I) and Sham 15Min (Sham-15). The tests performed will involve bioimpedance evaluation, blood lactate, electromyographic analysis and evaluation of maximum voluntary contraction by means of the maximal repetition test (1RM). Thus, the TLED will be applied on the muscle group to be evaluated, unilaterally, the same tests being repeated in the sequence. For analysis of the data, normality test will be used to verify the distribution and adequate statistical tests for the appropriate intra and intergroup comparisons, being considered two factors in the comparisons, time and group. A significance level of 5% will be adopted.

DETAILED DESCRIPTION:
It is a blinded randomized clinical trial. The athletes will undergo a previous evaluation (day 1) comprised by anamnesis and evaluation of the bioimpedance to analyze the body composition, will still carry out the evaluation of the load for a maximum repetition. Thus, 7 days after (day 2) the previous evaluation in the times immediately after and after 15 minutes of the LED application will be carried out new tests. These will involve assessment of blood lactate, heart rate variability and electromyography. In addition, during the execution of the fatigue protocol will be collected the number of repetitions of muscle contraction and its total execution time.

Due to the number of athletes that make up the university team (n = 19), cross-over will be necessary, where all athletes will initially be distributed to the 04 pre-defined groups in each subproject, and after the 7 days, they will be divided again.

ELIGIBILITY:
Inclusion Criteria:

* Handball practitioners;
* Absence of musculoskeletal injury in the last three months;
* Absence of anti-inflammatory and / or analgesic drugs 72 hours before the evaluations

Exclusion Criteria:

* Use of anabolic steroids;
* Presence of cardiovascular disease
* Use of alcohol and illicit drugs during the collection period

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-05-18 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Difference in number of repetitions | 2 years
  The present study was designed to detect the difference in the number of repetitions between the groups groups, after the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo RJ Guirro, Study Director — University of Sao Paulo
Locations (1):
- Universidade de São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The data will be shared in manuscript form

REFERENCES:
- [Result] Leal Junior EC, Lopes-Martins RA, Rossi RP, De Marchi T, Baroni BM, de Godoi V, Marcos RL, Ramos L, Bjordal JM. Effect of cluster multi-diode light emitting diode therapy (LEDT) on exercise-induced skeletal muscle fatigue and skeletal muscle recovery in humans. Lasers Surg Med. 2009 Oct;41(8):572-7. doi: 10.1002/lsm.20810. PMID 19731300
- [Result] Ferraresi C, Dos Santos RV, Marques G, Zangrande M, Leonaldo R, Hamblin MR, Bagnato VS, Parizotto NA. Light-emitting diode therapy (LEDT) before matches prevents increase in creatine kinase with a light dose response in volleyball players. Lasers Med Sci. 2015 May;30(4):1281-7. doi: 10.1007/s10103-015-1728-3. Epub 2015 Feb 27. PMID 25722067
- [Result] de Almeida P, Lopes-Martins RA, De Marchi T, Tomazoni SS, Albertini R, Correa JC, Rossi RP, Machado GP, da Silva DP, Bjordal JM, Leal Junior EC. Red (660 nm) and infrared (830 nm) low-level laser therapy in skeletal muscle fatigue in humans: what is better? Lasers Med Sci. 2012 Mar;27(2):453-8. doi: 10.1007/s10103-011-0957-3. Epub 2011 Jul 22. PMID 21814736